CLINICAL TRIAL: NCT07070882
Title: Effectiveness of an Oral Methylprednisolone Taper Following Primary Total Knee Arthroplasty
Brief Title: Oral Steroid Taper After Total Knee Arthroplasty
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Herbert John Cooper, MD, Associate Professor of Orthopedic Surgery, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAAV7426
Record Dates: First submitted 2025-06-28; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Patients receiving oral methylprednisolone (Experimental): Patients receiving a six-day oral methylprednisolone taper (21 tablets, 4 mg each) in addition to standard multimodal pain management
  Interventions: Drug: Methylprednisolone
- Patients receiving standard pain management without the taper (No Intervention): Patients receiving standard pain management without the taper

INTERVENTIONS:
Drug: Methylprednisolone — Patients will receive a tapered dose of methylprednisolone with the standard of care pain management
  Arms: Patients receiving oral methylprednisolone

SUMMARY:
This study aims to evaluate the effectiveness of an oral methylprednisolone taper in reducing postoperative pain, opioid consumption, and nausea following primary total knee arthroplasty (TKA).

DETAILED DESCRIPTION:
This study aims to evaluate the effectiveness of an oral methylprednisolone taper in reducing postoperative pain, opioid consumption, and nausea following primary total knee arthroplasty (TKA). While intravenous (IV) corticosteroids have been shown to provide short-term pain relief in the immediate postoperative period, their effects are limited to the first 24 hours. Given the inflammatory nature of TKA recovery, extending steroid administration through an oral taper may provide additional benefits in pain control, opioid reduction, and functional recovery. This study will assess whether adding an oral steroid taper to standard multimodal pain management improves clinical outcomes in TKA patients.This prospective, single-blinded, randomized controlled trial will enroll adults aged 18 and older undergoing primary TKA for osteoarthritis at Columbia University Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing primary TKA with a diagnosis of osteoarthritis
* > 18 years old
* Willingness to undergo randomization
* Patients who will be home by postoperative day (POD) #1 to start the dosing schedule that day (includes both ambulatory and POD #1 discharge patients)

Exclusion Criteria:

* Reported chronic corticosteroid or opiate use prior to surgery
* Prior Open Surgery on the Ipsilateral Knee
* Primary diagnosis other than osteoarthritis, including avascular necrosis, fracture, septic arthritis, or postoperative traumatic arthritis
* American Society of Anesthesiologists (ASA) score ≥ 4
* Reported history of liver disease, renal disease, or diabetes mellitus
* Current systemic fungal infection or other local infection
* Immunocompromised or immunosuppressed
* Current peptic ulcer disease
* History of psychosis, heart failure, myasthenia gravis, ocular herpes simplex virus, or systemic sclerosis
* Women with reported current pregnancy
* Known hypersensitivity to methylprednisolone
* ≤ 18 years old
* Inability to take oral medications
* Unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-06-20 (Estimated); Study Completion 2027-06-20 (Estimated)

PRIMARY OUTCOMES:
Surveys | Post-Operative Day 1, Day 2, Day 3, Day 4, Day 5, Day 6 Post-Operative 2-3 weeks, and Post-Operative 6-10 weeks
  Patient will report daily pain levels and nausea using Visual Analog Scale. The visual analog scale is from 0-10 with increments of 2 with 0 being no nausea and 10 being the worst and vomiting. Pain will also be documented similarly with 0 being no pain and 10 being the worst pain ever.

SECONDARY OUTCOMES:
Surveys | Post-Operative Day 1, Day 2, Day 3, Day 4, Day 5, Day 6 Post-Operative 2-3 weeks, and Post-Operative 6-10 weeks
  Patient will complete the KOOS Jr. Its calculates score from the survey questions answered with a score of 0 indicating knee disability and 100 representing perfect knee health.

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided